CLINICAL TRIAL: NCT06480565
Title: A Phase 1/2 Trial of ADI-270 (Engineered γδ Chimeric Receptor [CAR] Vδ1 T Cells Targeting CD70) in Adults With Relapsed or Refractory (R/R) Clear Cell Renal Cell Carcinoma (ccRCC)
Brief Title: A Phase 1/2 Trial of ADI-270 in ccRCC
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Adicet Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADI-202427001
Record Dates: First submitted 2024-06-25; First posted 2024-06-28 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: Renal cell carcinoma, cell therapy, CD70, chimeric antigen receptor (CAR) t-cell therapy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: 3+3 Dose Escalation Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation (Experimental): ADI-270 is administered at ascending dose levels as a single dose to determine the maximum tolerated dose (MTD) or maximum assessed dose (MAD) of ADI-270
  Interventions: Drug: ADI-270; Drug: Fludarabine; Drug: Cyclophosphamide
- Dose Expansion (Experimental): Dose Expansion with ADI-270 at the MTD/MAD to confirm recommended phase 2 dose (Part 2).
  Interventions: Drug: ADI-270; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: ADI-270 — Anti-CD70 CAR-T
Drug: Fludarabine — Chemotherapy for Lymphodepeletion
Drug: Cyclophosphamide — Chemotherapy for Lymphodepletion

SUMMARY:
This is a Phase 1/2 multicenter, open-label, dose escalation, and dose expansion study of ADI-270 - an Engineered gamma-delta Chimeric Receptor [CAR] Vδ1 T Cell product Targeting CD70 - in patients with R/R ccRCC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed clear cell RCC
2. Documented evidence of advanced or metastatic diseases.
3. Patients must have been treated with an immune checkpoint inhibitor and a VEGF inhibitor (the VEGF inhibitor must have been administered in the advanced and/or metastatic setting).
4. At least one measurable target lesion according to RECIST 1.1
5. At least three weeks, or 5 half-lives, whichever is shorter, from the last dose of the prior line of systemic therapy
6. KPS ≥ 70

Exclusion Criteria:

1. Subjects with CNS metastases or spinal cord compression are not eligible, unless they have completed therapy and have discontinued the use of corticosteroids for at least 8 weeks and remained stable prior to enrollment.
2. Clinically significant CNS dysfunction of any etiology in the opinion of the Investigator.
3. Prior radiation therapy within 21 days prior to start of study treatment with the exception of palliative radiotherapy to bone lesions (palliative radiotherapy to bone lesions must be completed at least 2 weeks prior to the first dose of LD).
4. Active malignancy (except for RCC, definitively treated basal or squamous cell carcinoma of the skin, and carcinoma in-situ of the cervix or bladder) within the past 24 months
5. Treatment with gene therapy, genetically modified cell therapy, or adoptive T cell therapy within 6 weeks before initiating LD in this study.
6. Receipt of CD70 targeted therapies for any indication
7. Require corticosteroid therapy > 5 mg per day of prednisone or equivalent.
8. History of any form of primary immunodeficiency such as severe combined immunodeficiency disease.
9. Presence of active autoimmune disease requiring ongoing systemic immunosuppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The Incidence of Subjects with Dose Limiting Toxicities within each dose level cohort | Day 28
  This primary endpoint will be used to determine the Maximum Tolerated Dose (MTD) or Maximum Assessed dose (MAD)
Proportion of treatment emergent and treatment related adverse events | 2 years
  This primary endpoint will be used to determine the MTD/MAD of ADI-270

CONTACTS AND LOCATIONS:
Locations (1):
- Adicet Clinical Trials, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nishimoto KP, Lamture G, Chanthery Y, Teague AG, Verma Y, Au M, Smith-Boeck M, Salum M, Murthy P, Gundurao SRY, Kaur R, Zhang J, Azameera A, Wong JTS, Speltz EB, Wang KM, Doan A, Sethuraman J, Bhatwala D, Giner-Rubio A, Puligujja P, Budworth H, Rold CJ, Panuganti S, Jakobovits A, Herrman M, Bhat A, Green S, Aftab BT. ADI-270: an armored allogeneic gamma delta T cell therapy designed to target CD70-expressing solid and hematologic malignancies. J Immunother Cancer. 2025 Jul 1;13(7):e011704. doi: 10.1136/jitc-2025-011704. PMID 40592738